CLINICAL TRIAL: NCT05381805
Title: Intensive (Pre)Clinical Characterization of Patients undergOing Atrial fibrillATion ablatlON: a Multicenter Clinical Care and Research Platform
Brief Title: ISOLATION 2.0: a Multicenter Clinical Care and Research Platform
Status: Not yet recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: NL80761.068.22
Record Dates: First submitted 2022-04-07; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
Keywords: Ablation; Pulmonary Vein Isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for analysis of circulating biomarkers of AF Possible biopts of the Left atrium in a subgroup of patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Treatment recommendations and guidelines for patients with atrial fibrillation (AF) are continuously changing. The role of catheter ablation in the treatment of AF increases and the techniques of the procedures are improving unceasingly. Responding to and evaluating the effect of these changes requires careful examination of this patient population and procedure outcomes. The aim is to create a clinical characterization platform for patients scheduled for AF ablations with the purpose to optimize health care processes and related translational research.

DETAILED DESCRIPTION:
Study design: Prospective cohort study and research platform of patients referred for AF ablation. Clinical characteristics and results of routine tests and procedures before, during and after AF ablation are collected. In addition, the following (non-standard) tests are performed: extended surface electrocardiogram (extECG), extended rhythm monitoring, biomarker testing, genetic analysis, and questionnaires. In subgroups of patients transesophageal electrocardiogram (TE-ECG), epicardial electroanatomical mapping and/or left atrial appendage (LAA) biopsy is performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Documented atrial fibrillation;
* Referred for any type of AF ablation: catheter ablation, stand-alone surgical AF ablation, surgical AF ablation concomitant with cardiac surgery, hybrid AF ablation, or redo AF ablation;
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Conditions preventing the patient from adhering from the study protocol;
* Emergency procedures.

A subject who meets any of the following criteria will be excluded from the subset in whom additional consent for transesophageal ECG-imaging is asked:

* Severe allergic reaction against contrast agents used in the CT- or MRI-protocol
* Severe allergic reaction against body surface electrodes

A subject who meets any of the following criteria will be excluded from the subset in whom additional consent for transesophageal ECG (TE-ECG) is asked:

• Status after esophageal or gastric surgery

A subject who meets any of the following criteria will be excluded from the subset in whom additional consent for Cardiovascular Magnetic Resonance (ISOLATION CMR) is asked:

• Contraindication to MRI

A subject who meets any of the following criteria will be excluded from the subset in whom additional consent for concomitant hybrid ablation of atrial fibrillation (COMBAT-AF) is asked:

• Prior catheter or surgical AF ablation.

Specific exclusion criteria for epicardial mapping (only applicable for patients undergoing hybrid or surgical AF ablation):

* Chronic obstructive pulmonary disease (COPD) Gold 11, 111, or IV;
* Heart failure, currently in New York Heart Association (NYHA) class Ill or IV;
* Any other pulmonary, cardiac, or other condition that may compromise a safe conduct of epicardial mapping in the opinion of the treating physician or investigator, taking the prolonged duration of single lung ventilation into account.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from two hospitals in the Netherlands with documented AF, referred for AF ablation.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Ablation success | 12 months
  Freedom from documented recurrence of atrial arrhythmia after 12 months. Recurrences in the first 3 months after the index procedure (blanking period) are exempted.

SECONDARY OUTCOMES:
Time to recurrence of AF or other atrial arrhythmia after the blanking period. | 3 to 24 months
  Time to recurrence of AF or other atrial arrhythmia after the blanking period of 3 months.
Early recurrences of AF or other atrial arrhythmia | 0 to 3 months
  Defined as any episode of documented arrhythmia during the blanking period, defined as within 3 months
Number of participants with disease progression to persistent or permanent AF. | 0 to 24 months
  Disease progression to persistent or permanent AF. Persistent AF is defined as AF that lasts longer than 7 days. Permanent AF can't be corrected with treatments.
Use of antiarrhythmic drugs (AADs) one year after ablation. | 0 to 24 months
  Use of antiarrhythmic drugs (AADs) one year after ablation
Interleukin 6 (IL-6) level | 0 to 24 months
  Change in circulating biomarker for substrate quantification.
Pro-brain natriuretic peptide 2 (pro-BNP2) level | 0 to 24 months
  Change in circulating biomarker for substrate quantification.
Fibroblast growth factor 23 (FGF-23) level | 0 to 24 months
  Change in circulating biomarker for substrate quantification.
Dickkopf-related protein 3 (DKK-3) level | 0 to 24 months
  Change in circulating biomarker for substrate quantification.
Angiopoietin 2 (ANG-2) level | 0 to 24 months
  Change in circulating biomarker for substrate quantification.
Endothelial cell-specific molecule 1 (ESM-1) level | 0 to 24 months
  Change in circulating biomarker for substrate quantification.
Insulin-like growth factor-binding protein 7 (IGFBP-7) level | 0 to 24 months
  Change in circulating biomarker for substrate quantification.
Bone morphogenetic protein 10 (BMP-10) level | 0 to 24 months
  Change in circulating biomarker for substrate quantification.
Redo procedures | 0 to 24 months
  Defined as repeated ablation procedure with the goal to prevent recurrence of AF or reduce the AF burden after one or more previous attempts to achieve the same goal.
Number of veins with pulmonary vein reconnection at redo procedure. | 0 to 24 months
  Number of veins with pulmonary vein reconnection at redo procedure.
Major adverse cardiovascular events (MACE). | 0 to 24 months
  Major adverse cardiovascular events (MACE).
Procedure time | Intraoperative
  Defined as skin-to-skin time (time from initial femoral vein puncture to time of removal of sheaths).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Vernooy, MD. PhD, Principal Investigator — Maastricht UMC+ & Radboudumc; Dominik Linz, MD, PhD, Principal Investigator — Maastricht UMC+ & Radboudumc & University of Adelaide and Royal Adelaide Hospital & University of Copenhagen; Ulrich Schotten, MD, PhD, Principal Investigator — Maastricht University & Cardiovascular Research Institute Maastricht